CLINICAL TRIAL: NCT03436927
Title: Comparison of the Effects of Two Different Virtual Reality Treatment Methods in Patients With Multiple Sclerosis: A Randomized Controlled Trial
Brief Title: Comparison of Two Different Virtual Reality Methods in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Yonca Zenginler, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YZenginler
Record Dates: First submitted 2017-12-11; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; rehabilitation; postural balance; exercise
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nintendo Wii Fit (Experimental): Participants in the Nintendo Wii group were included to exercise program that consisted of 16 individual PT-supervised sessions (two 60-minute sessions/week), which were prepared to improve balance. Each session started with 10 minutes of non-resistance cycling work for warm-up.
  Interventions: Other: Nintendo Wii Fit Balance exercises
- Balance Trainer (Experimental): Participants in the Balance Trainer group were included to exercise program that consisted of 16 individual PT-supervised sessions (two 60-minute sessions/week), which were prepared to improve balance. Each session started with 10 minutes of non-resistance cycling work for warm-up.
  Interventions: Other: Balance Trainer Balance Exercises
- Control (No Intervention): Patients in the 'Group III-control group' were included in the waiting list until the end of the study.

INTERVENTIONS:
Other: Nintendo Wii Fit Balance exercises — Nintendo Wii Fit' training protocol consisted of 'Penguin Slide', 'Table Tilt', 'Ski Slalom', 'Heading' and 'Balance Bubble' games that selected from the Wii Fit Plus balance games section
  Arms: Nintendo Wii Fit
Other: Balance Trainer Balance Exercises — Balance Trainer' training protocol consisted of 'Collect Apples', 'Outline', 'Paddle War' and 'Evaluation of Movement' games which were included in the device software and allowed the patients to done balance exercises in different directions.
  Arms: Balance Trainer

SUMMARY:
As a chronic, autoimmune, inflammatory disease of the central nervous system, Multiple Sclerosis (MS) is a neurologic problem which the most frequent cause of disability in young adults. Fatigue, pain, spasticity, muscle weakness, depression, as well as balance and gait disorders are amongst the symptoms of MS. Balance disorders and the falls caused by them are the most frequent problems which result in disability of MS patients, with 75% of all patients being affected during the course of disease. When considering previous studies carried out on physiotherapy and rehabilitation practices in the light of balance disorders and other related problems faced by MS patients, it can been that various physiotherapeutic approaches are applied with varying follow-up times and in the form of hospital sessions, home sessions, or group training. Posture and balance problems in MS patients are tried to be solved through long-lasting treatment sessions using traditional methods of physiotherapy, where less patient participation is observed. Fatigue, psychological impairment, and insufficient motivation are other aspects which influence the success of treatment and which need to be addressed in MS patients. In contrast to traditional methods of physiotherapy applied in form of long-lasting treatment sessions, technology-supported rehabilitation approaches have emerged in recent years. It can be seen that different systems have started to be employed in the physiotherapy of many chronic diseases, either alone or in company with traditional methods. Even though the clinical use of these systems is becoming widespread, there are certain gaps in terms of the systems' impacts, comparative advantages, or cost effectiveness. Keeping this in mind, the purpose of this study is to investigate and compare the impacts of 'Nintendo Wii Fit' and 'Balance Trainer', as two of the technologic methods with therapeutic impact which have started to be used for different diagnosis groups in recent years, on the balance and posture parameters of MS patients, with the ultimate aim to introduce a whole new point of view to traditional physiotherapy and rehabilitation studies.

ELIGIBILITY:
Inclusion Criteria:

* . Participants who were ambulatory and volunteer to participate to the study, in a stable phase of the disease, without relapses or worsening in the last 3 months, with an EDSS between 2.5-6 and aged between 25 to 60 years

Exclusion Criteria:

* physical activity more than 150 minutes per week, were pregnant, had blurred vision, had psychiatric problems, or severe cognitive impairment.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | Change between baseline and after 8 weeks of intervention were assessed.
  The Berg Balance Scale is a 56-point scale designed to measure balance among older people by the assessment of functional tasks. Its concurrent validity has been established for people with multiple sclerosis. The Berg Balance Scale is a five point ordinal scale and consisting of 14 balance activity. Each activity is scored between 0-4 and higher total scores indicating less impaired balance. 45-56=independent, 21-44=assisted walking, 0-20=dependent.

SECONDARY OUTCOMES:
Timed Up and Go Test | Change between baseline and after 8 weeks of intervention were assessed.
  The patient's mobility requiring both static and dynamic balance was assessed by Timed up and go test which measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again. A longer completion time indicates a higher risk of falling.
Six Minutes Walk Test | Change between baseline and after 8 weeks of intervention were assessed.
  Patients were instructed to walk a 30 m corridor for 6 minutes and the distance completed after 6 minutes (6MWD) was recorded.
Fatigue Severity Scale | Change between baseline and after 8 weeks of intervention were assessed.
  Fatigue severity scale is a nine-item, self-administered questionnaire that assesses the fatigue level in daily functions of MS patients. The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score=63. Higher fatigue severity scale scores indicating greater severity of fatigue.

IPD SHARING:
Plan to Share IPD: No